CLINICAL TRIAL: NCT06685991
Title: Effect of Timing of Dexamethasone Administration During Induction on Postoperative Outcomes: A Triple-Blinded Randomized Controlled Trial
Brief Title: Effect of Timing of Dexamethasone During Induction on Postoperative Outcomes
Acronym: TIDE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AABDI Mohammed (Other)
Collaborators: University Hospital Center Mohammed VI Tangier, Morocco (Unknown)
Responsible Party: Sponsor-Investigator, AABDI Mohammed, Assistant Professor of Anesthesiology and Critical Care, University Abdelmalek Essaadi faculty of medicine and pharmacy Tangier
Organization: University Abdelmalek Essaadi faculty of medicine and pharmacy Tangier (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHC M6 TANGIER
Record Dates: First submitted 2024-11-07; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Nausea and Vomiting (PONV); Postoperative Pain; Inflammatory Response to Wounding; Hyperglycemia Drug Induced; Hypotension on Induction; Timing of Dexamethasone Administration
Keywords: Dexamethasone; Timing of Administration; Anesthesia Induction; Randomized Controlled Trial (RCT); Triple-Blinded Study; Induction Protocol; Postoperative outcomes
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Participants in this study will be randomly assigned to one of three parallel groups to evaluate the effects of timing of dexamethasone administration during anesthesia induction on postoperative outcomes.
  Group 1 will receive dexamethasone before fentanyl administration. Group 2 will receive dexamethasone after the muscle relaxant administration. Group 3 (control) will receive no dexamethasone. This parallel assignment model allows for a direct comparison of outcomes across the three groups, examining factors such as postoperative nausea and vomiting, pain, glycemic control, and hemodynamic stability. Randomization and triple-blinding are implemented to minimize bias and improve the reliability of results.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study employs a triple-blinded design. Participants, care providers, investigators, and outcomes assessors are all blinded to the group assignments to prevent bias. Additionally, the study coordinators and data analysts responsible for interpreting results are also masked to maintain objectivity in data collection and analysis. Randomization is handled by an independent party, and group assignments are concealed until the completion of data analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexamethasone pre-induction (Experimental): Participants in this group will receive a single dose of dexamethasone administered intravenously before fentanyl administration during anesthesia induction. This arm assesses the impact of pre-fentanyl dexamethasone on postoperative outcomes, including nausea, pain, glycemic control, and hemodynamic stability.
  Interventions: Drug: Dexamethasone
- Dexamethasone post-induction (Experimental): Participants in this group will receive a single dose of dexamethasone administered intravenously after the muscle relaxant during anesthesia induction. This arm examines the effects of administering dexamethasone post-muscle relaxant on postoperative outcomes, including nausea, pain, glycemic control, and hemodynamic stability.
  Interventions: Drug: Dexamethasone
- No Dexamethasone (Control) (Placebo Comparator): Participants in this control group will not receive dexamethasone during anesthesia induction. This group serves as a baseline to compare the outcomes with those receiving dexamethasone at different timing points.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone will be administered intravenously at varying times during anesthesia induction to assess the impact of timing on postoperative outcomes. Participants will be randomized into one of three groups: one group will receive dexamethasone before the administration of fentanyl, a second group will receive it after the administration of a muscle relaxant, and a third control group will not receive dexamethasone. This timing variation aims to determine the optimal administration point to improve outcomes, including postoperative nausea, pain, glycemic stability, and hemodynamic response.

SUMMARY:
This study aims to investigate how the timing of dexamethasone administration during anesthesia induction affects patient outcomes after surgery. Dexamethasone is commonly used to reduce nausea and inflammation during and after surgery. However, it is not yet known if administering dexamethasone at different times during induction (before, during, or after specific anesthetic drugs) leads to better recovery and fewer postoperative complications.

Participants will be randomly assigned to one of three groups: one group will receive dexamethasone before fentanyl, another after the muscle relaxant, and a third group will not receive dexamethasone. This approach will help us understand if the timing of dexamethasone affects patient outcomes such as nausea, pain, and recovery quality. The study is triple-blinded, meaning that the participants, care providers, and investigators will not know which group the participants are in, to ensure unbiased results.

DETAILED DESCRIPTION:
This study explores the effects of different timings of dexamethasone administration during the induction phase of anesthesia on various postoperative outcomes. Dexamethasone is widely used in anesthesia practice to prevent postoperative nausea and vomiting (PONV) and to reduce inflammatory responses. However, the optimal timing of its administration has not been conclusively established, which may impact its effectiveness and patient recovery.

In this triple-blind randomized controlled trial, participants will be assigned to one of three intervention groups to receive dexamethasone at different times during anesthesia induction: (1) prior to fentanyl administration, (2) after administration of a muscle relaxant, or (3) no dexamethasone as a control group. We hypothesize that the timing of dexamethasone administration may influence outcomes such as incidence and severity of PONV, pain levels, time to recovery, and other potential complications.

By analyzing these parameters, the study seeks to establish an evidence-based guideline for the timing of dexamethasone administration to optimize postoperative recovery. The findings could inform anesthetic protocols and enhance patient outcomes in surgical settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Scheduled for elective non cardiac surgery requiring general anesthesia
* surgery last at least 90 minutes
* scare of more than 5 cm Able to provide informed consent Eligible for dexamethasone administration as part of routine perioperative care

Exclusion Criteria:

* Known allergy or hypersensitivity to dexamethasone or related corticosteroids
* History of uncontrolled diabetes mellitus or significant blood glucose management issues, as dexamethasone may affect glucose levels
* Severe cardiovascular instability or hemodynamic issues contraindicating study participation
* Patients receiving immunosuppressive therapy or with conditions affecting the immune system, as corticosteroids may alter immune responses
* Pregnancy or breastfeeding, due to potential risks to the fetus or infant
* Current or recent (within 30 days) use of other glucocorticoids, which may interfere with study outcomes
* Patients with psychiatric or cognitive conditions that impair their ability to consent or adhere to study protocols
* Lack of informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Nausea and Vomiting (PONV) | 24 hours
  To assess the frequency and severity of nausea and vomiting within the first 24 hours after surgery using APFEL scale

SECONDARY OUTCOMES:
Postoperative Pain Levels | At 2, 6, 12, and 24 hours postoperatively
  The Visual Analog Scale (VAS) ranges from 0 to 10, where 0 represents "no pain" and 10 represents "worst possible pain." Higher scores indicate greater pain intensity, representing a worse outcome.
Glycemic Variation before induction, 2 hours, and Immediate Postoperative Period | Baseline (immediately before induction), 2 hours after induction, and immediately after surgery
  Evaluate blood glucose levels at baseline Baseline (immediately before induction), 2 hours after induction, and immediately after surgery
Hypotension on Induction and during surgery | Record blood pressure at baseline (pre-induction), every 5 minutes during the induction period, and at the end of induction to evaluate stability.
  Record events of hypotension defined my mean arterial pressure (MAP) <65 mmHg or systolic arterial pressure (SAP) <90 mmHg or a drop by > 30% of baseline MAP or SAP.
Incidence of Postoperative Complications during first 24 postoperative hours | Up to 24 hours postoperatively
  Record any adverse events or complications that occur within the first 24 hours postoperatively, such as infections, respiratory issues, or other related complications.

IPD SHARING:
Plan to Share IPD: Undecided
Currently, there are no plans to share individual participant data (IPD) from this study due to considerations around patient privacy and data confidentiality. Given the sensitive nature of perioperative health data and the need to ensure participant anonymity, data sharing will only be considered if adequate safeguards can be implemented. Additionally, sharing IPD requires comprehensive agreements on data access, use, and security, which are not in place at this time.

REFERENCES:
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Wang JJ, Ho ST, Lee SC, Liu YC, Ho CM. The use of dexamethasone for preventing postoperative nausea and vomiting in females undergoing thyroidectomy: a dose-ranging study. Anesth Analg. 2000 Dec;91(6):1404-7. doi: 10.1097/00000539-200012000-00019. PMID 11093989